CLINICAL TRIAL: NCT04069546
Title: The Efficacy of Remote Ischemic Conditioning on Stroke-induced Immunodeficiency
Acronym: RIC-SIID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Clinical Professor, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RIC-SIID
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Remote ischemic preconditioning; Stroke-induced immunodeficiency; Stroke-associated Pneumonia; inflammation response
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIS-RIC (Experimental): RIC is a physical strategy performed through cuffs placed on the unilateral arm and inflated to 180 mmHg for 5-min followed by deflation for 5-min, the procedures are performed repeatedly for 5 times. This group of patients received regular therapy of acute ischemic stroke plus unilateral arm of RIC intervention.
  Interventions: Device: remote ischemic conditioning
- AIS (No Intervention): This group of patients received regular therapy of acute ischemic stroke.

INTERVENTIONS:
Device: remote ischemic conditioning — RIC is a physical strategy performed by an electric device with cuffs placed on the unilateral arm and inflated to 180 mmHg for 5-min followed by deflation for 5-min, the procedures are performed repeatedly for 5 times.
  Arms: AIS-RIC

SUMMARY:
to detect the effects of RIC on stroke-induced immunodeficiency and inflammation response in acute ischemic stroke patients

DETAILED DESCRIPTION:
Remote ischemic conditioning, consisting of several brief cycles of intermittent ischemia-reperfusion of the arm or leg, may potentially confer systemic protection against prolonged ischemia in a distant organ. Numerous reports have confirmed its strongest endogenous neuroprotection against brain injury after stroke, of which the immune mechanisms are majorly involved in RIC. At the same time, the inflammation response plays a great role in stroke development, which may expand the infarct area. Stroke-induced immunodeficiency can potentiate stroke-associated pneumonia, which is an important cause of death after strokes. In this study, the investigators will assess the effect of RIC on stroke-induced immunodeficiency and inflammation response in AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* Confirmed diagnosis of acute ischemic stroke(AIS) with onset of symptoms within 48h at recruitment;
* NIHSS score: ≤15;
* Prestroke modified Rankin Scale(mRS) ≤2;
* subject or his or her legally authorized representative was able to provide informed consent.

Exclusion Criteria:

* uncontrolled hypertension (defined as systolic blood pressure ≥200 mmHg);
* participation in another device or drug trial simultaneously;
* any vascular, soft tissue, or orthopedic injury (eg, superficial wounds and fractures of the arm) that contraindicated unilateral arm ischemic preconditioning;
* peripheral vascular disease (especially subclavian arterial and upper limb artery stenosis or occlusion);
* Women who have a positive pregnancy test;
* History of malignancies;
* Using remote ischemic conditioning within the preceding 1 week;
* known infection at admission;
* a history of infection or the use of antibiotics, immunosuppressants, or steroids within the preceding 3 months.
* Other conditions are not suitable for this trial (evaluated by researchers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-09-07 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
The changes of mHLA-DR level in plasma | change from baseline to 2(±24h)days, and at 7(±24h)days after admission
  through flow cytometry

SECONDARY OUTCOMES:
The changes of TLR-2, TLR-4 level in plasma | change from baseline to 2(±24h)days, and at 7(±24h)days after admission
  through flow cytometry
Incidence of Stroke-associated Pneumonia within 1 week | within 7(±24h)days after admission
  Stroke-associated Pneumonia diagnostic criteria base on the consensus of 2015
  Stroke-associated Pneumonia diagnostic criteria base on the consensus of 2015
  Stroke-associated Pneumonia diagnostic criteria base on the consensus of 2015
Number of Participants with physician-diagnosed pneumonia within 90 days after stroke onset | 90( ±7days) days after ischemic stroke onset
  Number of Participants with Physician-diagnosed Pneumonia within 90 days after stroke onset Physician-diagnosed Pneumonia within 90 days
White blood cell count, monocyte count | baseline, 2(±24h) days, 7(±24h) days after admission
  through routine blood test
Concentration of IL-1β、IL-6、IL-10、TNFα（CRP if patients are infected）level | baseline, 2(±24h)days, and at 7(±24h)days after admission
  inflammatory cytokines
Number of Participants with Favorable outcome at 90 days | 90 days after ischemic stroke onset
  definition of favorable outcome: mRS : 0-2 or NIHSS: 0-1
Number of Participants with any adverse events | during baseline to 90 days after stroke onset
  adverse events include stroke extension, gastrointestinal bleed, cardiac events, increased liver or renal enzymes, and transfer to intensive care unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, XI Cheng District,, China